CLINICAL TRIAL: NCT01887210
Title: A Pilot Gaming Adherence Program for Youth Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Dr. Larry K. Brown, Professor of Psychiatry and Human Behavior, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HD074846-01 (NIH)
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Adherence to HIV Treatment and Medication
Keywords: HIV; youth; medical adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMB Gaming Adherence Intervention (Experimental): Combination of smart pill bottle cap with mobile gaming application tailored for those living with HIV
  Interventions: Behavioral: IMB Gaming Adherence Intervention
- Enhanced treatment as usual (Active Comparator): Smart pill bottle cap and mobile phone but no game
  Interventions: Behavioral: Enhanced treatment as usual

INTERVENTIONS:
Behavioral: IMB Gaming Adherence Intervention — Combination of smart pill bottle cap with mobile gaming application tailored for those living with HIV
  Arms: IMB Gaming Adherence Intervention
Behavioral: Enhanced treatment as usual — Smart pill bottle cap and mobile phone but no game
  Arms: Enhanced treatment as usual

SUMMARY:
This study will develop and test a novel, technology based intervention to improve treatment adherence among youth living with HIV who are taking antiretroviral medication. In the intervention youth will access an engaging and immersive app/game on their smartphone.Data about the opening of the smart pill bottle will be transferred from the bottle cap wirelessly and will trigger a text message about their adherence. While gaming, participants will gain information about their health, improve motivation for ARV and medical appointment adherence, and practice healthy behaviors. If the Intervention is found to be effective, it can be tested in a larger study and then disseminated to other youth on antiretroviral medications.

DETAILED DESCRIPTION:
Despite need for consistent adherence to medical care, youth living with HIV (YLWH) have suboptimal rates of retention in care and adherence to antiretroviral medication (ARV) treatment. There are few adherence studies with YLWH and the results are mixed, so there is a great need for the development of novel interventions. Results of adult HIV adherence studies indicate that participants are interested in using technology-based methods and are most receptive toward interventions that couple technological devices with motivational components. Pill taking monitoring devices have been found to be a sensitive measure of adherence to ARV medications, but do not lead to sustained improvements in adherence or intrinsic motivation when used alone. Building on this knowledge, this study will examine a multi-level technology that integrates a medication monitoring device WITH an interactive smartphone based app/game that is attractive and engaging to YLWH. This multi-level approach will integrate theory driven content with novel, but intuitive, technology to improve HIV treatment adherence.

In this study, data on opening of the pill bottle will be transferred wirelessly from the bottle cap and a text on adherence sent to the phone. This developmental project will adapt and refine a smartphone app/game to include content consistent with the Information-Motivation-Behavioral Skills (IMB) Model. Creation and adaptation will occur from in-depth interviews with YLWH on ART (n=25) and an open trial of the Intervention (n=20). While gaming, participants will experience absorbing action-oriented adventures that increase information about their health (e.g. knowledge about HIV treatment), improve motivation (e.g. action-figures experience health benefits of adherence), and build skills (e.g. utilize clinicians as partners). A small randomized controlled pilot study (24 weeks) among 60 YLWH will examine the preliminary efficacy of the IMB Gaming Adherence Intervention (integration of the smart cap with the IMB informed app/game) compared to a comparison group who receive the smart cap and smartphone but no IMB game, on adherence and biological measures.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* in medical care for HIV and receiving antiretroviral treatment
* aware of their HIV status as per clinician and clinical record
* able to give consent/assent and not impaired by cognitive or medical limitations as per clinical assessment
* detectable viral load

Exclusion Criteria:

* none

Ages: 14 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-01-09 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry K Brown, MD, Principal Investigator — Rhode Island Hospital; Laura Whiteley, MD, Study Director — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Whiteley L, Brown L, Lally M, Heck N, van den Berg JJ. A Mobile Gaming Intervention to Increase Adherence to Antiretroviral Treatment for Youth Living With HIV: Development Guided by the Information, Motivation, and Behavioral Skills Model. JMIR Mhealth Uhealth. 2018 Apr 23;6(4):e96. doi: 10.2196/mhealth.8155. PMID 29685863

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IMB Gaming Adherence Intervention | Enhanced Treatment as Usual
Started | 33 | 33
Completed | 32 | 29
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes 61 participants. Participants that completed baseline and at least one follow-up assessment were included in the analytic sample.
Groups:
- Total: Total of all reporting groups
Arm/Group | IMB Gaming Adherence Intervention | Enhanced Treatment as Usual | Total
Number analyzed (Participants) | 32 | 29 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.5 (2.5) | 22.3 (2.5) | 22.4 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 25 | 23 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 32 | 29 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 28 | 59
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Started ARV in past 3 months [Count of Participants; unit: Participants]
  Yes | 11 | 11 | 22
  No | 21 | 18 | 39
Gaming Status [Count of Participants; unit: Participants] — Participants were asked about how often they played video games.
  Participants
    Daily or almost daily | 10 | 12 | 22
    Not everyday | 21 | 17 | 38
    Unknown or not reported | 1 | 0 | 1
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual | 9 | 7 | 16
  Homosexual | 17 | 18 | 35
  Bisexual | 5 | 2 | 7
  Undecided | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Log10 HIV-1 Viral Load
Description: Log viral load at end of study for participants with available viral load data (Log10 copies/ml)
Time Frame: 24 weeks
Population: Unable to extract viral load data from chart for 9 participants in IMB intervention and 1 in TAU+.
Measure: Mean (Standard Deviation); unit: Log10 copies/ml
Arm/Group | IMB Gaming Adherence Intervention | Enhanced Treatment as Usual
Number analyzed (Participants) | 23 | 28
Log10 copies/ml | 1.48 (2.07) | 1.82 (2.14)

2. Secondary Outcome: Electronically Measured Past 7-day Adherence
Description: Past 7 day medication adherence as measured by electronic medication monitoring device.
Time Frame: 24 weeks
Population: Missing data for n=1 from TAU+
Measure: Mean (Standard Deviation); unit: proportion of adherence
Arm/Group | IMB Gaming Adherence Intervention | Enhanced Treatment as Usual
Number analyzed (Participants) | 32 | 28
proportion of adherence | 0.29 (0.36) | 0.32 (0.36)

3. Secondary Outcome: Number of Kept Medical Appointments
Description: Number of kept medical appointments since baseline.
Time Frame: 24 weeks
Population: Unable to pull information from chart for 9 participants in the IMB intervention and 6 in the TAU+ groups.
Measure: Mean (Standard Deviation); unit: appointments kept since baseline
Arm/Group | IMB Gaming Adherence Intervention | Enhanced Treatment as Usual
Number analyzed (Participants) | 23 | 23
appointments kept since baseline | 1.78 (1.24) | 1.74 (1.32)

4. Other Pre Specified Outcome: Information-Motivation-Behavioral Skills (IMB) Antiretroviral Therapy (ART) Behavioral Skills Scale
Description: Behavioral Skills subscale from the Information-Motivation-Behavioral Skills (IMB) scale. This subscale measures self-efficacy for adherence to medical care related to antiretroviral medication and treatment. Five items were summed to get a total Behavioral Skills subscale score. Scores range from 5-25 where higher scores indicate greater self-efficacy for adherence to medical care related to ART medication and treatment.
Time Frame: 24 weeks
Population: Missing data for n=2 from IMB intervention, n=2 from TAU+
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IMB Gaming Adherence Intervention | Enhanced Treatment as Usual
Number analyzed (Participants) | 30 | 27
units on a scale | 19.83 (4.68) | 19.48 (5.12)

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Description: Adverse events as described in the study protocol were reported by study staff to the principle investigator.
Arm/Group | IMB Gaming Adherence Intervention | Enhanced Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

LIMITATIONS AND CAVEATS:
This study had a small sample. Participants were recruited from Jackson, MS, so this sample is not nationally representative. There is no perfect measure of adherence. Self-report and electronic monitoring devices assessments differed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No